CLINICAL TRIAL: NCT02241863
Title: The Effect of a Theory Based Educational Intervention on Medication Adherence to and Removes of Related Barriers in Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Head of the Social Determinants of Health Research Center, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 353
Record Dates: First submitted 2014-09-04; First posted 2014-09-16 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Patients With Bipolar Disorders
Keywords: bipolar disorders; medication adherence; psychological intervention; multifaceted intervention
MeSH Terms: conditions — Bipolar Disorder; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multifaceted intervention (Experimental): Patients, their caregivers and family members will received the educational and motivational interventions
  Interventions: Behavioral: Multifaceted intervention
- Active Comparator (Active Comparator): Usual Care The usual care group received routine counseling performed by the psychiatrist and nurses.
  Interventions: Behavioral: Routine counseling

INTERVENTIONS:
Behavioral: Multifaceted intervention — Supportive intervention: care giver, health care providers, and patient's family members (including disease knowledge, treatment t of the disease, medication problems or adverse effects, the importance of medication adherence, supervision taking medications by the patients as prescribed). patient education: about the disease and treatment, consuming regularly the pills motivational intervening, self-monitoring planning. Patients will attend in five motivational interviewing sessions regularly to facilitating and engaging intrinsic motivation within the patients in order to change medication adherence behavior.
  Arms: Multifaceted intervention
Behavioral: Routine counseling
  Arms: Active Comparator

SUMMARY:
Despite an increasing pharmacopoeia of effective medications for the treatment of bipolar disorder, patient outcomes continue to be impacted by treatment adherence. Non-adherence to treatments is also a major obstacle in translating efficacy in research settings into effectiveness in clinical practice. Non-adherence with bipolar disorder (BD) medication treatment dramatically worsens outcomes. Reasons for non-adherence among individuals with BD are multi-dimensional, and it has been suggested that a multifaceted intervention will be more effective. The study is aimed to assess the effectiveness of a multifaceted intervention on enhancing medications adherence in patients with bipolar disorders.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. meeting DSM-IV criteria for bipolar I or II disorder
3. concurrently treated with a mood stabilizer
4. not currently in weekly or biweekly psychotherapy
5. Persian speaking.

Exclusion Criteria:

* DSM-IV drug or alcohol misuse disorders (excluding nicotine),
* pregnancy or planning pregnancy in the next year
* requiring changing the drug or the dose of a mood stabilizer
* evidence of severe DSM-IV borderline personality
* Unable or unwilling to give written informed consent.
* An organic cerebral cause for bipolar disorder-for example, multiple sclerosis or stroke.
* intellectual disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
changes in Patient-reported medication Adherence to mood stabilizers | changes from baseline, 1 Months and 6 months follow-up
  The Medication Adherence Report Scale (MARS-5) will be used for assessing medication adherence to the mood stabilizers

SECONDARY OUTCOMES:
Plasma level of mood stabilizer | Changes from baseline, 1 Months and 6 months after the intervention
Changes in action planning | Changes from baseline, 1 Months and 6 months after the intervention
  A self-reported questionnaire on five 5-point scale that ranged from 1 (strongly disagree) to 5 (strongly agree)
Changes in coping planning | Changes from baseline, 1 Months and 6 months after the intervention
  A self-reported questionnaire on five 5-point scale that ranged from 1 (strongly disagree) to 5 (strongly agree)
Changes in quality of life | Changes from baseline, 1 Months and 6 months after the intervention
Changes in psychological predictors of medication adherence (intention, perceived behavioral control ,Self-monitoring and Behaviour Automaticity) | Changes from baseline, 1 Months and 6 months after the intervention
Changes in Global Impression for Bipolar Disorder Severity scale (CGI-BP-S) | Changes from baseline, 1 Months and 6 months after the intervention
Changes in Beliefs about Medicines Questionnaire (BMQ) | Changes from baseline, 1 Months and 6 months after the intervention
Changes in Young Mania Rating Scale (YMRS) | Changes from baseline, 1 Months and 6 months after the intervention
Changes in Montgomery Asberg Depression Rating Scale | Changes from baseline, 1 Months and 6 months after the intervention

CONTACTS AND LOCATIONS:
Locations (10):
- Iran (10):
  - Boostan, Ahvāz
  - Ebn'e Sina, Mashhad
  - 22 Bahman Hospital, Qazvin
  - Psychiatry Center, Semnan
  - Shahid Mahallati, Tabriz
  - Iran Psychiatry, Tehran
  - Maymanat, Tehran
  - Roozbeh, Tehran
  - Baharan, Zahedan
  - Dr. Beheshti, Zanjan

REFERENCES:
- [Derived] Pakpour AH, Modabbernia A, Lin CY, Saffari M, Ahmadzad Asl M, Webb TL. Promoting medication adherence among patients with bipolar disorder: a multicenter randomized controlled trial of a multifaceted intervention. Psychol Med. 2017 Oct;47(14):2528-2539. doi: 10.1017/S003329171700109X. Epub 2017 Apr 27. PMID 28446253